CLINICAL TRIAL: NCT06006819
Title: Plasma Proteomic Signature and the Prognosis of Acute Heart Failure With or Without Chronic Kidney Disease
Brief Title: Prognostic Markers of Acute Heart Failure With Chronic Kidney Disease
Status: Recruiting | Type: Observational
Sponsor: Cheng-Hsin General Hospital (Other)
Responsible Party: Principal Investigator, Shang Feng Yang, Physician, Cheng-Hsin General Hospital
Other Study IDs: CHGH(983)111A-61
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases; Acute Heart Failure; Biomarker
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute heart failure (AHF) is defined as new or worsening of symptoms and signs of heart failure and is the most frequent cause of unplanned hospital admission in elderly patients. N-terminal pro-brain natriuretic peptide (NT-pro-BNP) is one of the most developed prognostic markers for AHR patients and. NT-pro-BNP has limitations in terms of diagnostic or predictive accuracy in patients with chronic kidney disease (CKD). Plasma proteomics have the potential to examine underlying pathophysiological and prognostic roles, so we compared the plasma proteomic signature to predict outcomes of patients with or without CKD hospitalized for AHF.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized for acute heart failure

Exclusion Criteria:

* initial serum NT-proBNP level <300ng/ml, pregnancy, amputated, and end-stage renal disease under regular dialysis

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants were recruited from patients admitted to Cheng Hsin General Hospital with the major diagnosis of acute heart failure. After written informed consent was obtained (in compliance with the Helsinki Declaration), patients with age more than 20 were included. Exclusion criteria were initial serum NT-proBNP level <300ng/ml, the presence of amputation, being pregnant, and receiving regular dialysis.
Sampling Method: Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events | 1 year
  mortality, acute myocardial infarction, acute stroke, and heart failure hospitalization

SECONDARY OUTCOMES:
major adverse kidney events | 1 year
  mortality, new end-stage renal disease, and 30% decline in estimated GFR

CONTACTS AND LOCATIONS:
Overall Officials: Shang Feng Yang, MD, Principal Investigator — Cheng-Hsin General Hospital
Locations (1):
- Cheng Hsin General Hospital, Taipei, Baitou District, Taiwan